CLINICAL TRIAL: NCT00171626
Title: Efficacy and Safety of Diclofenac Sodium Gel in Knee Osteoarthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VOSG-PN-304
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2012-04-23 (Estimated); Status verified 2012-04

CONDITIONS: Osteoarthritis
Keywords: Knee osteoarthritis, Topical NSAID, Diclofenac sodium
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee

INTERVENTIONS:
Drug: Diclofenac Topical Sodium Gel 1%

SUMMARY:
This study will test the efficacy and safety of topical diclofenac sodium gel in the treatment of knee osteoarthritis.

ELIGIBILITY:
Key Inclusion criteria

* Osteoarthritis of the knee Key Exclusion criteria
* Other rheumatic disease, such as rheumatoid arthritis
* Active gastrointestinal ulcer during the last year
* Known allergy to analgesic drugs

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480
Dates: Start 2004-08; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
WOMAC pain score in target knee at Week 12
WOMAC physical function score in target knee at Week 12
Global rating of disease activity by patient at Week 12

SECONDARY OUTCOMES:
WOMAC pain and physical function scores in target knee and global rating of disease activity by patient at Weeks 1, 4 and 8
WOMAC stiffness score, pain on movement and spontaneous pain in target knee, and global rating of benefit by patient, at Weeks 1, 4, 8 and 12
Pain on movement in target knee and use of rescue medication recorded in diary
Global evaluation of treatment at final visit
Treatment responder rate according to OARSI criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Novartis Consumer Health Inc, Parsippany, New Jersey, United States

REFERENCES:
- [Derived] Baraf HS, Gloth FM, Barthel HR, Gold MS, Altman RD. Safety and efficacy of topical diclofenac sodium gel for knee osteoarthritis in elderly and younger patients: pooled data from three randomized, double-blind, parallel-group, placebo-controlled, multicentre trials. Drugs Aging. 2011 Jan 1;28(1):27-40. doi: 10.2165/11584880-000000000-00000. PMID 21174485